CLINICAL TRIAL: NCT05471973
Title: The Review and Improvement of Cardiac Implantable Device Infection Quality Initiative (RECTIFY) Demonstration Project
Brief Title: CIED Infection Quality Initiative Demonstration Project
Acronym: RECTIFY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Clinical Research Institute (Other); Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00110118
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Infections
Keywords: Cardiac Implantable Electronic Devices; Quality improvement
MeSH Terms: conditions — Infections | interventions — Patient Care Team; Weights and Measures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quality Improvement Program (Other): The quality improvement program will consist of development and/or refinement of participating health system's patient care pathways tailored to address the gaps and barriers around recognition and treatment of CIED infections. Interventions will be customized and modified as needed based on regular reviews and implementation progress.
  Interventions: Other: Multidisciplinary Team; Other: Outreach Visits; Other: Multifaceted Intervention; Other: Measurement and Feedback

INTERVENTIONS:
Other: Multidisciplinary Team — Multidisciplinary team will be established that will define gaps in care, monitor ongoing data, identify barriers to guideline-directed care, and develop and implement multifaceted intervention to address the barriers
Other: Outreach Visits — An outreach visit consulting group from the coordinating center and trial leadership will provide external guidance on reviewing data, defining barriers, and implementing interventions
Other: Multifaceted Intervention — These interventions are not limited to targeted engagement with non-extractors, electronic health record (EHR) decision support, creation of OR block time, use of opinion leaders, and development of clinical pathways. In addition, once patients are identified and referred to extraction centers, clinical pathways are needed to provide prompt care without clinical delay
Other: Measurement and Feedback — The coordinating center will provide ongoing feedback related to the site's data. This will include time to diagnosis, treatment, and outcomes related to the device infection.

SUMMARY:
The aim of this Quality Initiative (QI) demonstration project is to develop a model to increase guideline-driven care for patients with cardiovascular implantable electronic devices (CIED) infection. Multidisciplinary teams will be established to carry out the multifaceted intervention. This program seeks to improve early identification and diagnosis, appropriate treatment, and faster time to treatment of CIED infection.

DETAILED DESCRIPTION:
Retrospective data will be collected pre-intervention. The interventions will then be implemented for a total of six months and will continue through the data collection period. Prospective data collection will start three months after the intervention is started and will continue for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Cardiovascular Implantable Electronic Device (CIED) in place
* Presumed CIED infection, as defined by:

  1. Positive blood culture (two or more positive blood cultures for typical skin organisms (coagulase-negative staphylococci, Corynebacterium species, Propionobacterium species), or one positive blood culture for all other microorganisms), with no other source identified to explain the bacteremia
  2. Cases with definite evidence of pocket infection (defined as localized erythema, swelling, pain, tenderness, warmth, erosion, or drainage), if treated with antibiotics before culture, even with negative culture, will be considered device infection

Exclusion Criteria:

* Patients who are inappropriate for device extraction, for example those who are DNAR and not using therapy to prolong survival because any procedure is considered inappropriate and/or it is unlikely that extraction would change overall prognosis
* Death within one week of definitive CIED systemic infection diagnosis or positive blood culture. Cases of bacteremia originating from a source other than the CIED that resolve without any evidence of CIED involvement should not be considered as CIED infection
* Patients with left ventricular assist devices (LVADs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with CIEDs and positive blood cultures who receive extraction (per guidelines) | Up to 12 months
  Proportion of patients with CIEDs and positive blood cultures, who receive extraction
Proportion of patients with CIEDs and definite pocket infections who receive extraction (per guidelines) | Up to 12 months
  Proportion of patients with CIEDs and probable device infection, who receive extraction

SECONDARY OUTCOMES:
Proportion of patients with extraction within 7 days of diagnosis | Up to 12 months
  Proportion of patients who who receive extraction within 7 days and during index hospitalization
Proportion of patients with extraction during index hospitalization | Up to 12 months
Time from positive blood culture/clear pocket infection to extraction for those undergoing extraction | Up to 12 months
Number of patients identified with suspected CIED infection | Up to 12 months
Number of patients referred to both Extraction Center (from outside hospital) and electrophysiologists (at Extraction Center) for extraction | Up to 12 months
Number of actual extractions | Up to 12 months
Number of patients with multi-organ failure or septic shock at time of extraction | Up to 12 months
Estimated healthcare utilization/costs | Up to 12 months
Staff satisfaction as measured by a qualitative survey | Up to 12 months
Patient satisfaction as measured by a qualitative survey | Up to 12 months

OTHER OUTCOMES:
Mortality | Up to 12 months
  Number of deaths from CIED infection
Length of stay | Up to 12 months
  Clinical outcomes: number of days of hospitalization
Days of antibiotic treatments | Up to 12 months
  Number of days patient received antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Chris Granger, MD, Principal Investigator — Duke Clinical Research Institute; Sean Pokorney, MD, Principal Investigator — Duke Clinical Research Institute
Locations (3):
- United States (3):
  - Northwestern, Chicago, Illinois
  - Atrium Health, Charlotte, North Carolina
  - Moses Cone, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osude N, Granger CB, Young R, Al-Khalidil H, Ward K, Leyva M, Lambert C, Tillery M, Lin A, Mehta R, Satish M, Peigh G, Wright A, Epstein LM, Lundqvist CB, Piccini JP, Sohail MR, Pokorney SD. REview and improvement of cardiac implanTable device Infection management qualitY initiative (RECTIFY): Rationale and design for a cardiac implantable electronic device infection quality initiative demonstration project. Am Heart J. 2026 Feb;292:107264. doi: 10.1016/j.ahj.2025.08.017. Epub 2025 Aug 26. PMID 40876585